CLINICAL TRIAL: NCT05676463
Title: Phase 2 Study of Extreme Hypofractionation Including Pelvic Nodes for High Risk Prostate Cancer Using MgRT (MRI Guided Radiation Therapy)
Brief Title: MRI Guided Radiation Therapy for the Treatment of High Risk Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22D.687; JT 20770 (Other: JeffTrial Number)
Record Dates: First submitted 2022-12-13; First posted 2023-01-09 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Prostate Adenocarcinoma; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists; Glutamate Carboxypeptidase II; Magnetic Resonance Spectroscopy; X-Rays; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (MRI-guided IMRT, ADT) (Experimental): Patients undergo MRI-guided IMRT on study and receive SOC ADT throughout the trial. Patients may also undergo PSMA PET, CT, MRI, and bone scans at screening and undergo collection of blood samples throughout the trial.
  Interventions: Procedure: MRI-guided Intensity-Modulated Radiation Therapy; Drug: Antiandrogen Therapy; Procedure: PSMA PET Scan; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Bone Scan; Procedure: Biospecimen Collection; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: MRI-guided Intensity-Modulated Radiation Therapy — Undergo MRI-guided IMRT
Drug: Antiandrogen Therapy — Receive SOC ADT
  Other Names: ADT; Androgen Deprivation Therapy; Androgen Deprivation Therapy (ADT); Anti-androgen Therapy; Anti-androgen Treatment; Antiandrogen Treatment; Hormone Deprivation Therapy; Hormone-Deprivation Therapy
Procedure: PSMA PET Scan — Undergo PSMA PET scan
  Other Names: Prostate-specific Membrane Antigen PET; PSMA PET; PSMA-Positron emission tomography
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; computerized axial tomography; Computerized Tomography; CT; CT SCAN; tomography; Computerized axial tomography (procedure)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging; Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; nuclear magnetic resonance imaging; Magnetic resonance imaging (procedure)
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial tests whether magnetic resonance imaging (MRI)-guided hypofractionated radiation therapy works to reduce treatment time and side effects in patients with high risk prostate cancer. MRI-guided hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time directly to diseased tissue, reducing damage to healthy tissue. Using MRI-guided radiation therapy on areas of the prostate and pelvic lymph nodes may shorten overall treatment time compared to the longer standard of care therapy and may reduce the number and/or duration of side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate late grade 2+ genitourinary (GU) toxicity.

SECONDARY OBJECTIVE:

I. Evaluating acute GU and gastrointestinal (GI) toxicity, late GI toxicity, overall survival, prostate cancer specific survival, biochemical failure, and quality of life.

OUTLINE:

Patients undergo MRI-guided intensity-modulated radiation therapy (IMRT) on study and receive standard of care (SOC) antiandrogen therapy (ADT) throughout the trial. Patients may also undergo prostate specific membrane antigen (PSMA) positron emission tomography (PET), computed tomography (CT), MRI, and bone scans at screening and undergo collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for a total of 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Age: above 18 years
* Participants must be histologically proven, adenocarcinoma prostate
* Localized to the prostate without positive pelvic lymph node involvement
* No distant metastatic disease assessed by pretreatment PSMA PET or bone scan and CT scan
* High risk prostate cancer as defined by National Comprehensive Cancer Network (NCCN): Gleason score of 8- 10, clinical stage T3a or higher, or prostate specific antigen (PSA) > 20 ng/mL
* Ability to receive long term hormone therapy
* Karnofsky performance score (KPS) > 70
* No prior history of therapeutic irradiation to pelvis
* Patient willing and reliable for follow-up and quality of life (QOL)
* English speaking/reading

Exclusion Criteria:

* Evidence of distant or pelvic metastasis at any time since presentation
* Life expectancy < 2 years
* Previous radiation therapy (RT) to prostate or prostatectomy
* A previous trans-urethral resection of the prostate (TURP)
* Severe urinary symptoms or with severe International Prostate Symptom Score (IPSS) score despite being on hormonal therapy for 6 months which in the opinion of the physician precludes RT
* Patients with known obstructive symptoms with stricture
* Any contraindication to radiotherapy such as inflammatory bowel disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-11-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of late grade 2+ genitourinary (GU) toxicity | At 1 year
  Per Common Terminology Criteria for Adverse Events version 5.0 compared to rate of toxicity in POP-RT trial. Will be estimated for the entire sample that receives the intervention, treating death from any cause (other than treatment) as a competing risk and censoring subjects who drop out before experiencing toxicity at time of last follow-up. A point estimate of cumulative incidence at 1 year will be estimated from this curve along with a two-sided 90% confidence interval. If the upper bound of the interval is less than 20%, the null hypothesis will be rejected.

SECONDARY OUTCOMES:
Incidence of acute GU and gastrointestinal (GI) toxicity | At baseline
  Will be estimated using a binomial proportion and exact 95% confidence interval.
Incidence of acute GU and gastrointestinal (GI) toxicity | At treatment completion, up to 10 days
  Will be estimated using a binomial proportion and exact 95% confidence interval.
Incidence of acute GU and gastrointestinal (GI) toxicity | every 3 months after treatment until 1 year
  Will be estimated using a binomial proportion and exact 95% confidence interval.
Incidence of acute GU and gastrointestinal (GI) toxicity | every 6 months beginning at year 2, assessed up to 4 years
  Will be estimated using a binomial proportion and exact 95% confidence interval.
Incidence of late GI toxicity | At baseline
  Will be estimated using a binomial proportion and exact 95% confidence interval.
Incidence of late GI toxicity | At treatment completion, up to 10 days
  Will be estimated using a binomial proportion and exact 95% confidence interval.
Incidence of late GI toxicity | every 3 months after treatment until 1 year
  Will be estimated using a binomial proportion and exact 95% confidence interval.
Incidence of late GI toxicity | every 6 months beginning at year 2, assessed up to 4 years
  Will be estimated using a binomial proportion and exact 95% confidence interval.
Overall survival | At baseline
  Will be estimated using the Kaplan-Meier method.
Overall survival | At treatment completion, up to 10 days
  Will be estimated using the Kaplan-Meier method.
Overall survival | every 3 months after treatment until 1 year
  Will be estimated using the Kaplan-Meier method.
Overall survival | every 6 months beginning at year 2, assessed up to 4 years
  Will be estimated using the Kaplan-Meier method.
Prostate cancer specific survival | At baseline
  Will be estimated using the Kaplan-Meier method.
Prostate cancer specific survival | At treatment completion, up to 10 days
  Will be estimated using the Kaplan-Meier method.
Prostate cancer specific survival | every 3 months after treatment until 1 year
  Will be estimated using the Kaplan-Meier method.
Prostate cancer specific survival | every 6 months beginning at year 2, assessed up to 4 years
  Will be estimated using the Kaplan-Meier method.
Biochemical failure | At baseline
  Defined as prostate specific antigen nadir plus 2 ng/ml. Will be estimated using the Kaplan-Meier method.
Biochemical failure | At treatment completion, up to 10 days
  Defined as prostate specific antigen nadir plus 2 ng/ml. Will be estimated using the Kaplan-Meier method.
Biochemical failure | every 3 months after treatment until 1 year
  Defined as prostate specific antigen nadir plus 2 ng/ml. Will be estimated using the Kaplan-Meier method.
Biochemical failure | every 6 months beginning at year 2, assessed up to 4 years
  Defined as prostate specific antigen nadir plus 2 ng/ml. Will be estimated using the Kaplan-Meier method.
Quality of life measurement | At baseline
  Using patient reported outcome-expanded prostate cancer index composite. Will be summarized using descriptive statistics.
Quality of life measurement | At treatment completion, up to 10 days
  Using patient reported outcome-expanded prostate cancer index composite. Will be summarized using descriptive statistics.
Quality of life measurement | every 3 months after treatment until 1 year
  Using patient reported outcome-expanded prostate cancer index composite. Will be summarized using descriptive statistics.
Quality of life measurement | every 6 months beginning at year 2, assessed up to 4 years
  Using patient reported outcome-expanded prostate cancer index composite. Will be summarized using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Jessie DiNome, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States